CLINICAL TRIAL: NCT00958568
Title: A Study to Assess the Long-Term Efficacy and Safety of Olanzapine and Fluoxetine Combination Versus Fluoxetine Only in the Relapse Prevention of Stabilized Patients With Treatment-Resistant Depression
Brief Title: A Study in Relapse Prevention of Treatment-Resistant Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12115; H6P-MC-HDAY (Other: Eli Lilly and Company); CTRI/2009/091/000654 (Registry Identifier: Clinical Trials Register India)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — olanzapine-fluoxetine combination; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine and Fluoxetine combination (OFC) (Experimental)
  Interventions: Drug: Olanzapine and Fluoxetine combination (OFC)
- Fluoxetine (Active Comparator)
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Olanzapine and Fluoxetine combination (OFC) — Open label acute phase: introductory dose for 4 days then 3 milligram (mg) Olanzapine and 25 mg Fluoxetine Combination (3/25), 6/25, 12/25, 6/50, 12/50 or 18/50, oral, daily, for 6-8 weeks.
  Open label stabilization phase: 6/25, 12/25, 6/50, 12/50 or 18/50 mg, oral, daily for 16-20 weeks.
  Double blind relapse prevention phase: dose determined during stabilization phase at Week 17, oral, daily, for 27 weeks.
  Other Names: Symbyax; LY900000
  Arms: Olanzapine and Fluoxetine combination (OFC)
Drug: Fluoxetine — 25 or 50 mg/day fixed dosing for 27 weeks
  Other Names: Prozac; LY1101440
  Arms: Fluoxetine

SUMMARY:
The purpose of this study is to determine whether olanzapine and fluoxetine combination (OFC) if used for a long time (47 weeks) makes patients suffering from Treatment Resistant Depression stable, determine if OFC is safe when used to treat patients with Treatment Resistant Depression for a long time (up to 47 weeks), to determine whether olanzapine and fluoxetine combination or fluoxetine alone is better to treat Treatment Resistant Depression when treated for a long time (up to 47 weeks) and to assess the quality of life during treatment.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, active comparator-controlled, parallel study of participants with Treatment Resistant Depression (TRD), comparing the efficacy and safety of olanzapine and fluoxetine Combination (OFC) versus fluoxetine in relapse prevention of stabilized participants with TRD. The study will consist of 4 phases: a screening phase; a 6- to 8-week open-label acute treatment phase; a 10- to 12-week open-label stabilization phase; and a 27- to 29-week double-blind relapse prevention treatment phase. Participants who demonstrate response to open-label OFC during the acute treatment phase will continue into the stabilization phase. Participants who remain stable while receiving open-label OFC during this phase will be randomized to receive either OFC or fluoxetine during the double-blind relapse prevention phase. Investigators and participants will be blinded to the precise duration of the stabilization period, the definition of remission, and the criteria for entry into the relapse prevention phase; this information is described in a supplement given to Ethical Review Boards (ERBs) and regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

* Have single or recurrent unipolar Major Depressive Disorder (MDD), without psychotic features by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) clinical assessment, confirmed by the structured clinician Interview for DSM-IV Axis 1 disorders (SCID-I).
* If female and of childbearing potential, test negative for pregnancy and agree to abstain from sexual activity or use a medically accepted means of contraception during the study. Use of any oral or injectable contraception must be initiated prior to receiving treatment.
* Have 17-item Hamilton Depression (HAM-D) score greater than or equal to 18 at screening and the day treatment is due to be received for the first time.
* Have treatment-resistant depression, as defined by having demonstrated failure to achieve satisfactory antidepressant response to adequate separate treatment courses of at least 2 different antidepressants within the current episode of MDD.

Exclusion Criteria:

* Have a diagnosis of Parkinson's disease or related disorders.
* Have a current or lifetime diagnosis of any of the following according to DSM-IV criteria: Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, Psychotic Disorder Not Otherwise Specified, Bipolar Disorder I or II, Delirium of any type, Dementia of any type, Amnestic Disorder, any Substance-Induced Disorder, or any Psychotic Disorder due to a General Medical Condition.
* Have current diagnosis of post-partum depression, MDD with atypical features, or MDD with a seasonal pattern as defined in the DSM-IV.
* Have paranoid, schizoid, schizotypal, antisocial, and borderline personality disorders (Axis II) as a comorbid or primary diagnosis, based on DSM-IV criteria.
* Have had psychotic symptoms within 1 month prior to Screening or demonstrate psychotic features at screening and on the day treatment is due to be assigned for the first time as determined by the investigator.
* Have DSM-IV substance dependence/abuse or not willing to avoid use of the substance (not including dependence on nicotine or caffeine), as defined by the SCID-I, within the past 30 days.
* Are actively suicidal in the judgment of the investigator.
* Have had one or more seizures without a clear and resolved etiology.
* Have leukopenia or history of leukopenia without a clear and resolved etiology, or known history of agranulocytosis during the participant's lifetime.
* Have alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) values greater than or equal to 2 times the upper limit of normal (ULN) of the performing laboratory or aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) values greater than or equal to 2 times the ULN or total bilirubin values greater than or equal to 1.5 times the ULN at any time during screening.
* Have acute, serious, or unstable medical conditions.
* Have any illness such that death is anticipated within 1 year or intensive care unit hospitalization for the illness is anticipated within 6 months.
* Have elevated prolactin levels at screening.
* Have Bazett's corrected QT interval (QTc) greater than 450 milliseconds (male) or greater than 470 milliseconds (female) at screening and when treatment is due to be received for the first time.
* Have received electroconvulsive therapy (ECT) or vagus nerve stimulation (VNS) treatment within the current episode; have a history of failure to adequate treatment courses of ECT or VNS; or will require ECT or VNS at any time during study participation.
* If receiving psychotherapy, light therapy, or both, are anticipated to require changes in frequency/intensity of treatment regimen or to cease treatment regimen over the duration of the study. Participants who are not receiving any of these therapies upon study entry may not begin any of these therapies during screening, or during any treatment phases of the study.
* Have received previous treatment with clozapine.
* Have used a monoamine oxidase inhibitor (MAOI) within 14 days prior to screening or are expected to need MAOI treatment at any time during this study through 5 weeks after the participant discontinues from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (65):
- United States (36):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pasadena, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bridgeton, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Charles, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Kisco, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodstock, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellevue, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brown Deer, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Allis, Wisconsin
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banfield
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chennai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludhiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mysore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raipur
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Col. Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce, Puerto Rico
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khot'kovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nizhny Novgorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Village Nikolskoe
- South Africa (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Centurion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kempton Park
- Turkey (Türkiye) (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antalya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elâzığ
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gaziantep
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mersin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Şişli

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 4 treatment phases: a screening phase (Study Period I [SPI]) of 3 to 14 days; a 6- to 8-week (wk) acute open-label treatment phase (SPII); a 12-week open-label stabilization treatment phase (SPIII); and a 27-week double-blind (DB) randomized relapse prevention treatment phase (SPIV).
Groups:
- OFC (SPII ): Olanzapine and Fluoxetine Combination (OFC): 3 milligram (mg) Olanzapine and 25 mg Fluoxetine Combination (3/25), 6/25, 12/25, 6/50, 12/50 or 18/50, oral, daily, for 6-8 weeks during open-label acute treatment phase (SPII). Flexible dosing with initial forced titration.
- OFC (SPIII): 6 mg Olanzapine and 25 mg Fluoxetine Combination (OFC): 6 mg Olanzapine and 25 mg Fluoxetine Combination (6/25), 12/25, 6/50, 12/50 or 18/50 oral, daily, for 12 weeks during open-label stabilization treatment phase (SPIII). Flexible dosing.
- OFC (SPIV): Olanzapine and Fluoxetine Combination (OFC): 6 mg Olanzapine and 25 mg Fluoxetine Combination (6/25), 12/25, 6/50, 12/50 or 18/50, oral, daily, for 27 weeks during double-blind randomized relapse prevention treatment phase (SPIV). Fixed dosing.
- Flu (SPIV): Fluoxetine (Flu): 25 or 50 mg oral, daily, for 27 weeks during double-blind randomized relapse prevention treatment phase (SPIV).
Period: SPII (Wk 0-8, Acute Open-label)
Arm/Group | OFC (SPII ) | OFC (SPIII) | OFC (SPIV) | Flu (SPIV)
Started | 892 | 0 | 0 | 0
Completed | 655 | 0 | 0 | 0
Not Completed | 237 | 0 | 0 | 0
Not completed — Response Criteria Not Met | 80 | 0 | 0 | 0
Not completed — Adverse Event | 44 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 34 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 39 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0 | 0
Not completed — Protocol Violation | 13 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Sponsor Decision | 8 | 0 | 0 | 0
Not completed — Unknown, Not Otherwise Specified | 1 | 0 | 0 | 0
Period: SPIII (Wk 9-20,Open-label Stabilization)
Arm/Group | OFC (SPII ) | OFC (SPIII) | OFC (SPIV) | Flu (SPIV)
Started | 0 | 655 | 0 | 0
Completed | 0 | 444 | 0 | 0
Not Completed | 0 | 211 | 0 | 0
Not completed — Stabilization Criteria Not Met | 0 | 62 | 0 | 0
Not completed — Blinded Randomization Criteria Not Met | 0 | 30 | 0 | 0
Not completed — Adverse Event | 0 | 28 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 41 | 0 | 0
Not completed — Protocol Violation | 0 | 24 | 0 | 0
Not completed — Lost to Follow-up | 0 | 9 | 0 | 0
Not completed — Entry Criteria Not Met | 0 | 6 | 0 | 0
Not completed — Sponsor Decision | 0 | 5 | 0 | 0
Not completed — Physician Decision | 0 | 4 | 0 | 0
Not completed — Relapse Criteria Met | 0 | 1 | 0 | 0
Not completed — Unknown, Not Otherwise Specified | 0 | 1 | 0 | 0
Period: SPIV (Wk 21-47, DB Relapse Prevention)
Arm/Group | OFC (SPII ) | OFC (SPIII) | OFC (SPIV) | Flu (SPIV)
Started | 0 | 0 | 221 | 223
Completed | 0 | 0 | 139 | 117
Not Completed | 0 | 0 | 82 | 106
Not completed — Relapse Criteria Met | 0 | 0 | 24 | 63
Not completed — Adverse Event | 0 | 0 | 19 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 16 | 15
Not completed — Protocol Violation | 0 | 0 | 11 | 5
Not completed — Lost to Follow-up | 0 | 0 | 3 | 8
Not completed — Sponsor Decision | 0 | 0 | 5 | 4
Not completed — Entry Criteria Not Met | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- OFC (SPII-Wk 0-8, Acute Open-label): Olanzapine and Fluoxetine Combination (OFC): 3 milligram (mg) Olanzapine and 25 mg Fluoxetine Combination (3/25), 6/25, 12/25, 6/50, 12/50 or 18/50, oral, daily, for 6-8 weeks during open-label acute treatment phase (SPII). Flexible dosing with initial forced titration.
Arm/Group | OFC (SPII-Wk 0-8, Acute Open-label)
Number analyzed (Participants) | 892
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.38 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 591
  Male | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 167
  Not Hispanic or Latino | 725
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27
  Asian | 115
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 101
  White | 634
  More than one race | 11
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 533
  Mexico | 44
  Puerto Rico | 20
  Argentina | 53
  Turkey | 28
  Russian Federation | 66
  South Africa | 40
  India | 108
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m²)] — N=892, data was not reported for 1 participant
  kilograms/square meter (kg/m²) | 29.12 (7.36)

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse by Any Criteria
Description: Relapse defined as meeting any of these criteria: 50% increase in Montgomery-Asberg Depression Rating Scale (MADRS) score from randomization with a Clinical Global Impressions-Severity (CGI-S) of Depression score increase to a score of 4 or more; Hospitalized for depression or suicidality; Discontinued due to lack of efficacy/worsening of depression/suicidality. MADRS is a 10-item rating scale for depressive mood symptoms severity, items rated on 0-6 scale, with total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (the most extremely ill). Lack of Efficacy/Worsening of depression was at discretion of investigator based on clinical observation. Suicidality is thoughts or actions of self-harm as determined by the investigator. Those who did not relapse were "censored" at their last observation.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants are included in the time to event analyses. The numbers of participants censored are 186 and 152 for OFC and Flu groups, respectively.
Measure: Median (Full Range); unit: days
Groups:
- OFC (SPIV): Olanzapine and Fluoxetine Combination (OFC): 6 milligram (mg) Olanzapine and 25 mg Fluoxetine Combination (6/25), 12/25, 6/50, 12/50 or 18/50, oral, daily, for 27 weeks during double-blind randomized relapse prevention treatment phase (SPIV).
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
days | NA (10.0) [6.0 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion. | NA (5.9) [7.0 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion.
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Power estimate assumes approximately 1230 participants enter SPII. With a 60% drop-out/disqualification rate in SPII, then 492 participants enter SPIII. If 26% of participants drop out during SPIII, then 364 participants enter SPIV. Assuming 20% drop-out rate, 25% relapse rate on OFC and 40% relapse rate for fluoxetine (hazard ratio = 0.56), the log-rank test is 80% powered to detect a difference at a 2-sided 0.05 level. A total of 95 relapse events during SPIV should satisfy these assumptions; Test type: Superiority or Other; p < 0.001, Log Rank — The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons

2. Secondary Outcome: Percentage of Participants Who Relapse by Any Criteria
Description: Relapse is defined as meeting any of the following criteria: 50% increase in Montgomery-Asberg Depression Rating Scale (MADRS) score from randomization with concomitant Clinical Global Impressions-Severity (CGI-S) of Depression score increase to a score of 4 or more; Hospitalization for depression or suicidality; Discontinuation due to lack of efficacy/worsening of depression/suicidality. MADRS is a rating scale for severity of depressive mood symptoms with 10 items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (the most extremely ill). Lack of Efficacy/Worsening of depression was at the discretion of the investigator and based on clinical observation. Suicidality is thoughts or actions of self-harm as determined by the investigator.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants | 15.8 | 31.8
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Relapse rates were analyzed using the Cochran-Mantel-Haenszel test adjusting for country

3. Secondary Outcome: Percentage of Participants Who Relapse Based on Montgomery-Åsberg Depression Rating Scale (MADRS) Score With Concomitant Clinical Global Impressions-Severity (CGI-S) of Depression Score
Description: Relapse is defined as a 50% increase in the Montgomery-Asberg Depression Rating Scale (MADRS) score from randomization with concomitant Clinical Global Impressions-Severity (CGI-S) of Depression score increase to a score of 4 or more. The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (the most extremely ill).
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants | 14.0 | 28.3
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Relapse rates were analyzed using the Cochran-Mantel-Haenszel test adjusting for country

4. Secondary Outcome: Percentage of Participants Who Relapse as Measured by Hospitalization for Depression or Suicidality
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants | 1.8 | 1.3
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.713, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Relapse rates were analyzed using the Cochran-Mantel-Haenszel test adjusting for country

5. Secondary Outcome: Percentage of Participants Who Relapse as Measured by Discontinuation Due to Lack of Efficacy/Worsening of Depression/Suicidality
Description: Lack of Efficacy/Worsening of depression was at the discretion of the investigator and was based on clinical observation. Suicidality is thoughts or actions of self-harm as determined by the investigator.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants | 10.9 | 28.3
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Relapse rates were analyzed using the Cochran-Mantel-Haenszel test adjusting for country

6. Secondary Outcome: Time to Relapse Based on the Montgomery-Åsberg Depression Rating Scale (MADRS) Score With Concomitant Clinical Global Impressions-Severity (CGI-S) of Depression Score
Description: Relapse is defined as a 50% increase in the Montgomery-Asberg Depression Rating Scale (MADRS) score from randomization with concomitant Clinical Global Impressions-Severity (CGI-S) of Depression score increase to a score of 4 or more. The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (the most extremely ill). Those who did not relapse were "censored" at their last observation.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants are included in the time to event analyses. The numbers of participants censored are 190 and 160 for OFC and Flu groups, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
days | NA (10.4) [6 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion. | NA (6.2) [7 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion.
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Time to Relapse as Measured by Hospitalization for Depression or Suicidality
Description: Those who did not relapse were "censored" at their last observation.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants are included in the time to event analyses. The numbers of participants censored are 217 and 220 for OFC and Flu groups, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
days | NA (29.9) [6 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion. | NA (4.3) [7 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion.
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.831, Log Rank — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to Relapse as Measured by Discontinuation Due to Lack of Efficacy/Worsening of Depression/Suicidality
Description: Lack of Efficacy/Worsening of depression was at the discretion of the investigator and was based on clinical observation. Suicidality is thoughts or actions of self-harm as determined by the investigator. Those who did not relapse were "censored" at their last observation.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants are included in the time to event analyses. The numbers of participants censored are 197 and 160 for OFC and Flu groups, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
days | NA (11.8) [6 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion. | NA (5.3) [7 to NA] — Not calculable due to few participants reaching the time-to-event endpoint of relapse at study completion.
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of Participants Responding to Treatment During Open-Label Acute Treatment Phase
Description: A 50% or greater improvement from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS) and a Clinical Global Impressions-Severity (CGI-S) of Depression score ≤3 will be considered as response criteria met. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Week 0 to Week 8
Population: All participants who entered open-label acute treatment phase (SPII).
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPII-Wk 0-8, Acute Open-label)
Number analyzed (Participants) | 892
percentage of participants | 78.0

10. Secondary Outcome: Percentage of Participants Maintaining Response at Any Point During Stabilization Treatment Phase
Description: as for outcome 9
Time Frame: Week 8 to Week 20
Population: All participants who entered open-label stabilization treatment phase (SPIII).
Measure: Number; unit: percentage of participants
Groups:
- OFC (SPIII): Olanzapine and Fluoxetine Combination (OFC): 6 mg Olanzapine and 25 mg Fluoxetine Combination (6/25), 12/25, 6/50, 12/50 or 18/50 oral, daily, for 12 weeks during open-label stabilization treatment phase (SPIII). Flexible dosing.
Arm/Group | OFC (SPIII)
Number analyzed (Participants) | 655
percentage of participants | 68.2

11. Secondary Outcome: Percentage of Participants Achieving Remission at Any Point During Stabilization Treatment Phase
Description: Remission is defined as the Montgomery-Asberg Depression Rating Scale (MADRS) score ≤8. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Week 8 to Week 20
Population: All participants who entered open-label stabilization treatment phase (SPIII).
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIII)
Number analyzed (Participants) | 655
percentage of participants | 77.9

12. Secondary Outcome: Percentage of Participants Maintaining Remission
Description: as for outcome 11
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants | 86.4 | 78.9
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Remission rates were analyzed using the Cochran-Mantel-Haenszel test adjusting for country

13. Secondary Outcome: Mean Change From Week 20 to Week 47 in Montgomery-Asberg Depression Rating Scale (MADRS) Using Mixed-Effects Model Repeated Measures (MMRM) Analysis
Description: The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) Mean values were controlled for baseline (Week 20), treatment, country, visit, and treatment by visit interaction.
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) MADRS measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 221
units on a scale | 2.06 (0.56) | 4.97 (0.61)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -2.91, 95% CI 2-sided [-4.46 to -1.36], Standard Error of Mean 0.78

14. Secondary Outcome: Mean Change From Week 20 to Week 47 in Montgomery-Asberg Depression Rating Scale (MADRS) Using Last Observation Carried Forward (LOCF) Analysis
Description: The MADRS has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) Mean values were controlled for baseline (Week 20), treatment and country.
Time Frame: Randomization (Week 20), up to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) MADRS measurements. LOCF principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 221
units on a scale | 3.03 (0.71) | 6.84 (0.73)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment and country; LS Mean Difference = -3.82, 95% CI 2-sided [-5.39 to -2.24]

15. Secondary Outcome: Mean Change From Week 20 to Week 47 in Clinical Global Impressions - Severity (CGI-S) of Depression Using Mixed-Effects Model Repeated Measures (MMRM) Analysis
Description: CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) Mean values were controlled for baseline (Week 20), treatment, country, visit, and treatment by visit interaction.
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) CGI-S measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 221
units on a scale | 0.20 (0.08) | 0.54 (0.08)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.002, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -0.34, 95% CI 2-sided [-0.55 to -0.12], Standard Error of Mean 0.11

16. Secondary Outcome: Resource Utilization - Average Number of Hours Worked for Pay Per Week at Week 47
Time Frame: Week 47
Population: All randomized participants who worked for pay at Week 47.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 70 | 63
hours | 37.49 (16.95) | 37.76 (14.58)

17. Secondary Outcome: Resource Utilization (Number of Psychiatric Visits, Number of Emergency Room or Equivalent Facility Visits for Psychiatric Illness)
Description: Resource utilization is defined as the average number of psychiatric visits and number of emergency room or equivalent facility visits for psychiatric illness.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who provided information of psychiatric visits and emergency room or equivalent facility visits for psychiatric illness from Week 21 to Week 47.
Measure: Mean (Standard Deviation); unit: visits per participant
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 138 | 115
visits per participant
  Psychiatric visits (n=136, 113) | 0.65 (1.43) | 0.81 (1.52)
  Emergency room or equivalent facility visits | 0.00 (0.00) | 0.00 (0.00)

18. Secondary Outcome: Change From Week 20 to Week 47 Endpoint in the Sheehan Disability Scale (SDS)
Description: The SDS is completed by the participant and is used to assess the effect of the participant's symptoms on their work or school (Item 1), social (Item 2), and family life and home responsibilities (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Total scores is the sum of the 3 items and range from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Least Squares (LS) Mean values were controlled for baseline (Week 20), treatment and country.
Time Frame: Randomization (Week 20), up to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) SDS score measurements. Last observation carried forward (LOCF) principle was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 154 | 167
units on a scale | 1.30 (0.72) | 3.24 (0.73)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.007, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment and country; LS Mean Difference = -1.94, 95% CI 2-sided [-3.36 to -0.53], Standard Error of Mean 0.72

19. Secondary Outcome: Percent of Participants With Treatment-Emergent Akathisia
Description: Barnes Akathisia Scale (BAS) rates observable, restless movements of drug-induced akathisia as well as the subjective awareness of restlessness and any distress associated with the akathisia. It consists of 4 items. 3 items (objective akathisia, subjective awareness of restlessness and subjective distress related to restlessness) rated on a 4-point scale, with 0 being no akathisia and 3 being severe akathisia. Item 4 (global clinical assessment of Akathisia) is derived from the responses on Items 1-3 rated on a 6-point scale, with 0 being absence and 5 being extreme Akathisia. Treatment emergent akathisia is defined as a global clinical assessment score on BAS <2 at baseline (Week 20) and a global clinical assessment score on BAS ≥2 post-baseline (Weeks 21-47).
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) BAS measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 217 | 213
percentage of participants | 0.9 | 0.9
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Percent of Participants With Treatment-Emergent Parkinsonism
Description: Simpson-Angus Scale is used to measure Parkinsonian-type symptoms in participants exposed to neuroleptics. The scale consists of 10 items, each rated on a 5-point scale, with 0 meaning complete absence of the condition and 4 meaning the presence of the condition in extreme form. The total score is obtained by adding the items and ranges from 0-40 with higher scores indicating worse conditions. Treatment emergent parkinsonism is defined as total score ≤3 of items 1 through 10 of the Simpson-Angus scale at baseline (Week 20) and a total score >3 of items 1 through 10 post-baseline (Weeks 21-47).
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) Simpson-Angus Scale measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 214 | 208
percentage of participants | 1.4 | 0.0
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.248, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

21. Secondary Outcome: Percent of Participants With Treatment-Emergent Dyskinesia
Description: Abnormal Involuntary Movement Scale (AIMS) is a 12-item scale designed to record the occurrence of dyskinetic movements. Items 1 through 10 are rated on a 5-point scale, with 0 being no dyskinetic movements and 4 being severe dyskinetic movements. Items 11 and 12 are yes/no questions regarding the dental condition of the participants. Treatment emergent dyskinesia is defined as a score ≥3 on any one of the AIMS items 1-7 post-baseline (Weeks 21-47) or scores ≥2 on any two of the AIMS items 1-7 post-baseline (Weeks 21-47) among participants without either criteria at baseline (Week 20).
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) AIMS measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 212 | 208
percentage of participants | 0.5 | 0.0
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

22. Secondary Outcome: Mean Change From Week 20 to Week 47 in Fasting Total Cholesterol
Description: Mixed-effects model repeated measures (MMRM) analysis was used to calculate Least Squares (LS) Mean and standard error (SE). LS Mean values were controlled for baseline (Week 20), treatment, country, visit, and treatment by visit interaction.
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) cholesterol measurements.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 212 | 209
milligrams/deciliter (mg/dL) | -2.65 (3.24) | -1.74 (3.52)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.839, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -0.91, 95% CI 2-sided [-9.71 to 7.89], Standard Error of Mean 4.47

23. Secondary Outcome: Percent of Participants With Treatment-Emergent High Fasting Total Cholesterol
Description: Borderline to High fasting total cholesterol: ≥200 milligrams/deciliter (mg/dL) and <240 mg/dL at baseline and ≥240 mg/dL any time post baseline; Normal to Borderline fasting total cholesterol: <200 mg/dL at baseline, ≥200 mg/dL and <240 mg/dL any time post baseline; Normal to High fasting total cholesterol: <200 mg/dL at baseline and ≥240 mg/dL any time post baseline.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had borderline or normal cholesterol level at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) cholesterol measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 75 | 83
percentage of participants
  Borderline to High (n= 75, 83) | 28.0 | 20.5
  Normal to Borderline (n=47, 59) | 17.0 | 16.9
  Normal to High (n=47, 59) | 2.1 | 3.4
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.352, Fisher Exact — P-value is for Borderline to High. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value is for Normal to Borderline. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — P-value is for Normal to High. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons

24. Secondary Outcome: Mean Change From Week 20 to Week 47 in Fasting Low-Density Lipoprotein (LDL) Cholesterol
Description: as for outcome 22
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) LDL cholesterol measurements.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 200 | 203
milligrams/deciliter (mg/dL) | -0.72 (2.96) | 0.85 (3.20)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.703, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -1.57, 95% CI 2-sided [-9.69 to 6.54], Standard Error of Mean 4.12

25. Secondary Outcome: Percent of Participants With Treatment-Emergent High Fasting Low-Density Lipoprotein (LDL) Cholesterol
Description: Borderline to High fasting LDL cholesterol: ≥100 milligrams/deciliter (mg/dL) and <160 mg/dL at baseline and ≥160 mg/dL any time post baseline; Normal to Borderline fasting LDL cholesterol: <100 mg/dL at baseline, ≥100 mg/dL and <160 mg/dL any time post baseline; Normal to High fasting LDL cholesterol: <100 mg/dL at baseline and ≥160 mg/dL any time post baseline.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had borderline or normal LDL cholesterol value at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) LDL cholesterol measurements.
Measure: Number; unit: percent of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 115 | 134
percent of participants
  Borderline to High (n= 115, 134) | 17.4 | 10.4
  Normal to Borderline (n=22, 26) | 22.7 | 30.8
  Normal to High (n=22, 26) | 4.5 | 0.0
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.139, Fisher Exact — [p-value comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.746, Fisher Exact — [p-value comment as in outcome 23, analysis 2]
Statistical Analysis 3: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.458, Fisher Exact — [p-value comment as in outcome 23, analysis 3]

26. Secondary Outcome: Mean Change From Week 20 to Week 47 in Fasting High-Density Lipoprotein (HDL) Cholesterol
Description: as for outcome 22
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) HDL cholesterol measurements.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 211 | 207
milligrams/deciliter (mg/dL) | -1.71 (0.84) | 2.02 (0.92)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -3.73, 95% CI 2-sided [-5.99 to -1.47], Standard Error of Mean 1.15

27. Secondary Outcome: Percent of Participants With Treatment-Emergent Low Fasting High-Density Lipoprotein (HDL) Cholesterol
Description: Normal to Low fasting HDL cholesterol is ≥40 milligrams/deciliter (mg/dL) at baseline and <40 mg/dL anytime post baseline.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had normal HDL cholesterol value at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) HDL cholesterol measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 199 | 208
percentage of participants | 39.2 | 25.5
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.004, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

28. Secondary Outcome: Percent of Participants With Treatment-Emergent Hepatic Events
Description: Participants with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3 times the upper limit of normal (ULN) at baseline, with ALT or AST >=3 times the ULN post-baseline and total bilirubin >=2 times ULN at the same time are considered having treatment-emergent hepatic events.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had baseline (Week 20) and post-baseline (Weeks 21-47) hepatic function measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 209 | 208
percentage of participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

29. Secondary Outcome: Mean Change From Week 20 to Week 47 in Fasting Triglycerides
Description: as for outcome 22
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) triglycerides measurement.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 211 | 209
milligrams/deciliter (mg/dL) | -8.24 (5.70) | -21.51 (6.20)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.083, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = 13.27, 95% CI 2-sided [-1.72 to 28.26], Standard Error of Mean 7.62

30. Secondary Outcome: Percent of Participants With Treatment-Emergent High Fasting Triglycerides
Description: Borderline to High fasting triglycerides: ≥150 milligrams/deciliter (mg/dL) and <200 mg/dL at baseline and ≥200 mg/dL any time post baseline; Normal to Borderline fasting triglycerides: <150 mg/dL at baseline, ≥150 mg/dL and <200 mg/dL any time post baseline; Normal to High fasting triglycerides: <150 mg/dL at baseline and ≥200 mg/dL any time post baseline.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had borderline or normal triglycerides value at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) triglyceride measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 68 | 74
percentage of participants
  Borderline to High (n=47, 41) | 51.1 | 26.8
  Normal to Borderline (n= 68, 74) | 22.1 | 6.8
  Normal to High (n=68, 74) | 16.2 | 5.4
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.029, Fisher Exact — [p-value comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.014, Fisher Exact — [p-value comment as in outcome 23, analysis 2]
Statistical Analysis 3: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.054, Fisher Exact — [p-value comment as in outcome 23, analysis 3]

31. Secondary Outcome: Mean Change From Week 20 to Week 47 in Fasting Glucose
Description: as for outcome 22
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) glucose measurements.
Measure: Least Squares Mean (Standard Error); unit: milligrams/deciliter (mg/dL)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 200 | 198
milligrams/deciliter (mg/dL) | 3.67 (1.36) | -2.22 (1.47)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.002, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = 5.89, 95% CI 2-sided [2.22 to 9.56], Standard Error of Mean 1.87

32. Secondary Outcome: Percent of Participants With Treatment-Emergent High Fasting Glucose
Description: Impaired to High fasting glucose: ≥100 milligrams/deciliter (mg/dL) and <126 mg/dL at baseline and ≥126 mg/dL any time post baseline; Normal to High glucose: <100 mg/dL at baseline and ≥126 mg/dL any time post baseline; Normal to Impaired fasting glucose is <100 mg/dL at baseline, ≥100 mg/dL and <126 mg/dL any time post baseline; Normal/Impaired to High fasting glucose: <126 mg/dL at baseline and ≥126 mg/dL any time post baseline.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had impaired or normal glucose value at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) glucose measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 188 | 193
percentage of participants
  Impaired to High (n=98, 97) | 18.4 | 7.2
  Normal to High (n=90, 96) | 4.4 | 5.2
  Normal to Impaired (n=90, 96) | 35.6 | 28.1
  Normal/Impaired to High (n= 188, 193) | 11.7 | 6.2
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.031, Fisher Exact — P-value is for Impaired to High. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 1.00, Fisher Exact — [p-value comment as in outcome 23, analysis 3]
Statistical Analysis 3: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.344, Fisher Exact — P-value is for Normal to Impaired. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons
Statistical Analysis 4: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.072, Fisher Exact — P-value is for Normal/Impaired to High. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons

33. Secondary Outcome: Mean Change From Week 20 to Week 47 in Weight
Description: as for outcome 22
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) weight measurements.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 222
kilograms (kg) | 1.14 (0.33) | -2.78 (0.36)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = 3.92, 95% CI 2-sided [2.96 to 4.88], Standard Error of Mean 0.49

34. Secondary Outcome: Percent of Participants With Week 20-to-Week 47 Endpoint Increase in Weight of at Least 7%
Time Frame: Week 20 to Week 47
Population: All randomized participants who had Week 20 and at least 1 post-baseline (Weeks 21-47) weight measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 222
percentage of participants | 11.8 | 2.3
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p < 0.001, Fisher Exact — The threshold for statistical significance was 0.05

35. Secondary Outcome: Percent of Participants With Suicide-Related Thoughts and Behaviors
Description: Columbia Suicide Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) C-SSRS measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 220 | 221
percentage of participants
  Suicidal Ideation | 4.1 | 6.3
  Suicidal Behavior | 0 | 0
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.392, Fisher Exact — P-value is for suicidal ideation. The test was run using an a priori 2-sided threshold for statistical significance of 0.05. No adjustments were made for multiple comparisons

36. Secondary Outcome: Mean Change in Corrected (for Rate) Cardiac QT Interval Using Fridericia's Formula (QTcF) on Electrocardiogram
Description: Least Squares (LS) Mean values were obtained from a mixed model repeated measures (MMRM) analysis. Model includes baseline (Week 20), treatment, country, visit, and treatment by visit interaction.
Time Frame: Randomization (Week 20), Week 47
Population: All randomized participants who had baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) electrocardiogram (ECG) measurements.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 201 | 194
milliseconds (msec) | -3.12 (1.48) | -1.55 (1.60)
Statistical Analysis 1: Comparison: OFC (SPIV) vs Flu (SPIV); Test type: Superiority or Other; p = 0.421, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; The model adjusted for baseline (Week 20), treatment, country, visit, and treatment-by-visit interaction; LS Mean Difference = -1.57, 95% CI 2-sided [-5.42 to 2.27], Standard Error of Mean 1.95

37. Secondary Outcome: Percent of Participants With Treatment-Emergent Corrected (for Rate) Cardiac QT Interval Using Fridericia's Formula (QTcF) on Electrocardiogram ≥500 Milliseconds (Msec)
Description: Data presented are the percent of participants whose baseline corrected (for rate) cardiac QT interval <500 msec with post-baseline corrected (for rate) cardiac QT interval ≥500 msec.
Time Frame: Randomization (Week 20) to Week 47
Population: All randomized participants who had <500 msec QTc interval at baseline (Week 20) and at least 1 post-baseline (Weeks 21-47) electrocardiogram (ECG) measurements.
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 214 | 214
percentage of participants | 0 | 0

38. Secondary Outcome: Percent of Participants With a 60 Milliseconds (Msec) Increase in Fridericia-Corrected (for Rate) Cardiac QT Interval (QTcF) on Electrocardiogram
Time Frame: Randomization (Week 20) to Week 47
Population: as for outcome 36
Measure: Number; unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 214 | 214
percentage of participants | 0 | 0

39. Other Pre Specified Outcome: Kaplan-Meier Estimate of Percentage of Subjects Not Relapsing at Week 27 (Day 189)
Description: Relapse is defined as meeting any of the following criteria (Relapse-any reason): 50% increase in MADRS score from randomization with concomitant CGI-S of Depression score increase to a score of 4 or more (MADRS score/CGI-S Depression Score); Hospitalization for depression or suicidality; Discontinuation due to lack of efficacy/worsening of depression/suicidality. MADRS is a rating scale for severity of depressive mood symptoms with 10 items rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). CGI-S measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (the most extremely ill). Lack of Efficacy/Worsening of depression was at the discretion of the investigator and based on clinical observation. Suicidality is thoughts or actions of self-harm as determined by the investigator.
Time Frame: Randomization (Week 20) to Week 27
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OFC (SPIV) | Flu (SPIV)
Number analyzed (Participants) | 221 | 223
percentage of participants
  Relapse-any criteria | 83.6 [77.6 to 88.1] | 66.5 [59.6 to 72.5]
  Relapse-MADRS score/CGI-S Depression Score | 85.3 [79.3 to 89.6] | 69.6 [62.7 to 75.5]
  Relapse-Hospitalization for depression/suicidality | 97.7 [94.0 to 99.1] | 98.6 [95.6 to 99.5]
  Relapse-Discontinued for lack efficacy/worsening | 87.4 [81.7 to 91.4] | 69.8 [63.0 to 75.6]

ADVERSE EVENTS:
Groups:
- OFC (SPII): Olanzapine and Fluoxetine Combination (OFC): 3 milligram (mg) Olanzapine and 25 mg Fluoxetine Combination (3/25), 6/25, 12/25, 6/50, 12/50 or 18/50, oral, daily, for 6-8 weeks during open-label acute treatment phase (SPII). Flexible dosing with initial forced titration.
Arm/Group | OFC (SPII) | OFC (SPIII) | OFC (SPIV) | Flu (SPIV)
Serious Adverse Events (participants affected / at risk) | 13/892 | 9/655 | 9/221 | 7/223
Other Adverse Events (participants affected / at risk) | 606/892 | 348/655 | 100/221 | 105/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OFC (SPII) (N=892) | OFC (SPIII) (N=655) | OFC (SPIV) (N=221) | Flu (SPIV) (N=223)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event resulted in death
Headache (Nervous system disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | OFC (SPII) (N=892) | OFC (SPIII) (N=655) | OFC (SPIV) (N=221) | Flu (SPIV) (N=223)
Constipation (Gastrointestinal disorders) | 24 (25) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 20 (20) | 5 (5) | 5 (5) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 125 (129) | 8 (8) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 15 (17) | 7 (7) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 34 (37) | 18 (19) | 10 (10) | 8 (9)
Vomiting (Gastrointestinal disorders) | 12 (12) | 15 (15) | 6 (6) | 4 (5)
Fatigue (General disorders) | 68 (74) | 15 (15) | 2 (2) | 2 (2)
Irritability (General disorders) | 12 (12) | 2 (2) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 32 (34) | 11 (12) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (5) | 9 (9) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 9 (9) | 10 (12) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 6 (6) | 6 (7) | 3 (3)
Influenza (Infections and infestations) | 8 (8) | 12 (12) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 37 (40) | 23 (23) | 9 (12) | 12 (13)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 20 (20) | 11 (22) | 7 (9)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Blood glucose increased (Investigations) | 9 (10) | 4 (4) | 4 (4) | 1 (1)
Blood prolactin increased (Investigations) | 0 (0) | 12 (12) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 17 (18) | 15 (15) | 4 (4) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Weight increased (Investigations) | 151 (155) | 59 (60) | 8 (8) | 5 (5)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 1 (1) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 123 (129) | 11 (11) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 6 (7) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 9 (9) | 3 (3) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 4 (4)
Akathisia (Nervous system disorders) | 12 (12) | 9 (9) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 13 (13) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 29 (31) | 6 (6) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 64 (76) | 39 (55) | 15 (60) | 13 (24)
Hypersomnia (Nervous system disorders) | 12 (12) | 6 (6) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 10 (10) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 9 (9) | 1 (1) | 1 (1) | 1 (1)
Sedation (Nervous system disorders) | 61 (66) | 17 (20) | 3 (5) | 0 (0)
Somnolence (Nervous system disorders) | 76 (82) | 20 (21) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 33 (34) | 10 (11) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 21 (23) | 12 (12) | 2 (2) | 9 (9)
Depression (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2) | 12 (12)
Initial insomnia (Psychiatric disorders) | 10 (18) | 7 (8) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 20 (24) | 16 (17) | 8 (11) | 16 (26)
Libido decreased (Psychiatric disorders) | 14 (14) | 6 (6) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 22 (24) | 7 (7) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1/78 (1) | 0/70 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (9) | 5 (5) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days